CLINICAL TRIAL: NCT02872051
Title: Integrated Mental Health Care and Vocational Rehabilitation to Individuals on Sick Leave Due to Anxiety and Depression in Denmark (the Danish IBBIS Study): A Multi-center Randomized Controlled Trial
Brief Title: Integrated Mental Health Care and Vocational Rehabilitation to Individuals on Sick Leave Due to Anxiety and Depression
Acronym: IBBIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amager Hospital (Other)
Collaborators: The Danish Agency for Labour Market and Recruitment (Other); Copenhagen Municipality, Denmark (Other Government); Gentofte Municipality, Denmark (Unknown); Municipality of Lyngby-Taarbæk, Denmark (Unknown); Gladsaxe Municipality, Denmark (Other)
Responsible Party: Principal Investigator, Lene Falgaard Eplov, MD, PhD, Amager Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IBBIS Anxiety Depression
Record Dates: First submitted 2016-08-15; First posted 2016-08-18 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Generalized Anxiety; Social Phobia; Panic Disorder; Depression
Keywords: Vocational Rehabilitation; Anxiety; Depression; Common Mental Disorders; Cognitive Behavior Therapy; Return to Work; Mental Health Services; Integration
MeSH Terms: conditions — Generalized Anxiety Disorder; Phobia, Social; Panic Disorder; Depression; Anxiety Disorders | interventions — Rehabilitation, Vocational

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Standard treatment and standard vocational rehabilitation
- IBBIS MHC (Experimental): IBBIS mental health care and standard vocational rehabilitation
  Interventions: Behavioral: IBBIS mental health care and standard vocational rehabilitation
- IBBIS integrated MCH and VR (Experimental): Integrated mental health care and vocational rehabilitation
  Interventions: Other: Integrated mental health care and vocational rehabilitation

INTERVENTIONS:
Behavioral: IBBIS mental health care and standard vocational rehabilitation — Standard vocational rehabilitation.
  Stepped mental health care provided by the IBBIS mental health care team (e.g. nurses, psychologists, and medical doctors) with the treatment modalities:
  Psychoeducation Bibliotherapy Cognitive-behavior Therapy Monitoring and reassessment
  Arms: IBBIS MHC
Other: Integrated mental health care and vocational rehabilitation — Integrated mental health care and vocational rehabilitation provided by the IBBIS team. The IBBIS team is composed by employment specialists from the municipal job centers and health care professionals from the mental health services (e.g. nurses, psychologists, and medical doctors).
  Mental health care is provided according to a stepped care model with the following treatment modalities:
  Psychoeducation Bibliotherapy Cognitive-behavior Therapy Monitoring and reassessment
  Vocational rehabilitation is inspired by Individual Placement and Support and is a workplace-oriented intervention with problem-solving conversations as a core element
  Arms: IBBIS integrated MCH and VR

SUMMARY:
The purpose of this study is to investigate the efficacy of 1) a stepped mental health care intervention and 2) an integrated mental health care and vocational rehabilitation intervention for people on sick leave because of depression and anxiety in Denmark

DETAILED DESCRIPTION:
Background:

Depression and anxiety are important contributors to the global burden of disease and causes negative effects on both the individual and society. Depression and anxiety are very likely to influence the individual's workability and up to 40 % of the people on sick leave in Denmark have common mental disorders like depression and anxiety. There is no clear evidence that mental health care alone will provide sufficient support for vocational recovery for this target group. Integrated vocational and health care services have shown good effects on return to work in other Scandinavian countries.

Objective:

The purpose of the Danish IBBIS study is to examine the efficacy of 1) a stepped mental health care intervention and 2) an integrated mental health care and vocational rehabilitation intervention for people on sick leave because of depression and anxiety in Denmark.

Method:

This three-arm, randomized, controlled trial is set up to investigate the effectiveness of the stepped mental health care model and the integrated mental health care and vocational rehabilitation intervention for people on sick leave because of depression and anxiety in Denmark. 603 patients are recruited from Danish job centers in four municipalities. The primary outcome is return to work at 12 months.

Results/discussion:

This study will contribute with new knowledge on vocational recovery and integrated vocational and health care interventions in a Scandinavian context.

ELIGIBILITY:
Inclusion Criteria:

* Depression, Generalized Anxiety, Social Phobia or Panic Disorder according to Mini International Neuropsychiatric Interview (MINI)
* On sick leave from work or unemployment and have received sick leave benefit for minimum four weeks OR have started a sick leave benefit case which is estimated to last for minimum eight weeks
* Citizen in one of the following municipalities: Copenhagen City, Gladsaxe Municipality, Lyngby-Taarbæk Municipality or Gentofte Municipality
* Danish-speaking
* Given informed consent

Exclusion Criteria:

* Pregnant
* High degree of suicidal ideation
* Dementia
* Alcohol or substance misuse that hinders the person participating in treatment
* Wish to start or continue psychological therapy
* Need for psychiatric treatment in the secondary psychiatric care system
* Medically unstable to a degree that the patient cannot adhere to treatment
* Participant in the research project Collabri
* Attending stress courses in the stress clinics of Copenhagen City
* Assessed by job center case managers to be dangerous

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 631 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Time to return to work | 12 months
  Time from baseline to first return to work for more than four consecutive weeks

SECONDARY OUTCOMES:
Work | 12 months
  Competitive work 12 months after baseline (yes/no)
Time to return to work | 24 months
  Time from baseline to first return to work for more than four consecutive weeks
Recurrent Sickness Absence | 24 months
  Time from baseline to recurrent sickness absence for more than 8 weeks
Degree of depressive symptoms | 6 months
  Self-assessed depressive symptoms by the Beck Depression Inventory (BDI)
Degree of anxiety symptoms | 6 months
  Self-assessed anxiety symptoms by the Beck Anxiety Inventory (BAI)
Degree of psychological stress symptoms | 6 months
  Self-assessed psychological stress by the Cohen perceived stress scale (PSS)
Work and social functioning | 6 months
  Work and social functioning by the Work and Social Adjustment Scale (WSAS)

OTHER OUTCOMES:
Symptom level | 6, 12 and 24 months
  Symptom level on de four dimensions: Distress, Depression, Anxiety and Somatization by 4-dimensional symptom questionnaire (4DSQ)
Death | 6, 12 and 24 months
  Death and cause of death by register data
Suicidal ideation | 6, 12 and 24 months
  Suicidal ideation by BDI
Life-threatening conditions | 6, 12 and 24 months
  Life-threatening conditions by register data

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Services of the Capital Region of Denmark, Copenhagen, Capital Region of Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hoff A, Poulsen RM, Fisker JP, Hjorthoj C, Nordentoft M, Christensen U, Bojesen AB, Eplov LF. Integrated Mental Healthcare and Vocational Rehabilitation for People on Sick Leave with Anxiety or Depression: 24-Month Follow-up of the Randomized IBBIS Trial. J Occup Rehabil. 2023 Sep;33(3):570-580. doi: 10.1007/s10926-023-10094-7. Epub 2023 Feb 27. PMID 36849841
- [Derived] Hoff A, Poulsen RM, Fisker J, Hjorthoj C, Rosenberg N, Nordentoft M, Bojesen AB, Eplov LF. Integrating vocational rehabilitation and mental healthcare to improve the return-to-work process for people on sick leave with depression or anxiety: results from a three-arm, parallel randomised trial. Occup Environ Med. 2022 Feb;79(2):134-142. doi: 10.1136/oemed-2021-107894. Epub 2021 Dec 16. PMID 34916330
- [Derived] Poulsen R, Hoff A, Fisker J, Hjorthoj C, Eplov LF. Integrated mental health care and vocational rehabilitation to improve return to work rates for people on sick leave because of depression and anxiety (the Danish IBBIS trial): study protocol for a randomized controlled trial. Trials. 2017 Dec 2;18(1):578. doi: 10.1186/s13063-017-2272-1. PMID 29197414

DOCUMENTS (2):
  • Study Protocol (2019-07-05): https://cdn.clinicaltrials.gov/large-docs/51/NCT02872051/Prot_001.pdf
  • Statistical Analysis Plan (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT02872051/SAP_002.pdf